CLINICAL TRIAL: NCT06748729
Title: Investigation on Performance of a New Developed Prosthetic Knee
Brief Title: Clinical Investigation (Beta) of a New Developed Prosthetic Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP2023120529
Record Dates: First submitted 2024-04-17; First posted 2024-12-27 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Amputation
Keywords: Trans-femoral; Prosthetic knee; Amputees

STUDY DESIGN:
Intervention Model Description: The test will be a non-randomized single group repeated measures open label prospective design with observational and self-report measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Exploratory testing of a new prosthetic knee (Experimental): The investigational device is provided to subjects, who then use it as their main prosthesis for a period of 4 weeks prior to returning for data collection on the device.
  Interventions: Device: Navii Knee

INTERVENTIONS:
Device: Navii Knee — Microprocessor controlled prosthetic knee (MPK)

SUMMARY:
The aim of this investigation is to evaluate the efficacy of the investigational device regarding performance improvements and satisfaction in descending activities for moderate to high active prosthesis users within the intended population for the investigational device. Additionally, the overall satisfaction for activities of daily living will be evaluated after a certain time of use (4 weeks home use).

DETAILED DESCRIPTION:
This investigation is a non-randomized single group repeated measures open label prospective design with observational and self-report measures.

Two scheduled study events are planned for amputee subjects, with 4 weeks between visits.

ELIGIBILITY:
Inclusion Criteria:

* 45Kg< body weight < 136Kg
* Cognitive ability to understand all instructions and questionnaires in the study;
* Unilateral TF/KD amputees that are regular prosthesis users for at least 3 months
* Current MPK users (passive MPKs only) regularly performing descent activities (stairs/ramps)
* Age ≥ 18 years
* Willing and able to participate in the study and follow the protocol

Exclusion Criteria:

* Users with stump pain
* Users with socket problems
* Pregnant Users
* Users using Power Knee, Kenevo or mechanical knees as their prescribed prosthesis
* Alignment that cannot be matched with the Navii setup, as described in Instructions for use.
* Osseointegration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt N. Gruben, Principal Investigator — Össur Americas
Locations (1):
- Össur Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 11 subjects were enrolled, but only 10 completed the protocol and were included in the data analysis.
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Amputation level Transfemoral [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction on Ramp Descent With the New Microprocessor-controlled Prosthetic Knee (MPK)
Description: Satisfaction on ramp descent with the new MPK compared to prescribed device In-house questionnaire and Scale used: worse, same, better.
Time Frame: After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Count of Participants; unit: Participants
Groups:
- Exploratory Testing of a New Prosthetic Knee: New Microprocessor controlled prosthetic knee (MPK)
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
Participants
  Rheo Knee Users: number analyzed (Participants) | 4
  Rheo Knee Users: worse | 1
  Rheo Knee Users: same | 0
  Rheo Knee Users: better | 3
  Hydraulic Users: number analyzed (Participants) | 6
  Hydraulic Users: worse | 4
  Hydraulic Users: same | 1
  Hydraulic Users: better | 1

2. Primary Outcome: Satisfaction on Stair Descent With the New Microprocessor-controlled Prosthetic Knee (MPK)
Description: Satisfaction on stair descent with the new MPK compared to prescribed device In-house questionnaire and Scale used: worse, same, better
Time Frame: After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Count of Participants; unit: Participants
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
Participants
  In-house questionnaire Rheo Knee Users: number analyzed (Participants) | 4
  In-house questionnaire Rheo Knee Users: worse | 0
  In-house questionnaire Rheo Knee Users: same | 1
  In-house questionnaire Rheo Knee Users: better | 3
  In-house questionnaire Hydraulic Users: number analyzed (Participants) | 6
  In-house questionnaire Hydraulic Users: worse | 5
  In-house questionnaire Hydraulic Users: same | 0
  In-house questionnaire Hydraulic Users: better | 1

3. Primary Outcome: Satisfaction on Level Ground Walking Activity
Description: Satisfaction on level ground walking activity with the new MPK compared to prescribed device In-house questionnaire and Scale used: worse, same, better
Time Frame: After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Count of Participants; unit: Participants
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
Participants
  Rheo Knee users: number analyzed (Participants) | 4
  Rheo Knee users: Worse | 0
  Rheo Knee users: Same | 4
  Rheo Knee users: Better | 0
  Hydraulic users: number analyzed (Participants) | 6
  Hydraulic users: Worse | 0
  Hydraulic users: Same | 6
  Hydraulic users: Better | 0

4. Primary Outcome: Change in Overall Satisfaction From Baseline With Prescribed Device to After 4 Weeks of Investigational Device Use
Description: The PEQ (Prosthesis Evaluation Questionnaire) assesses the quality of life and satisfaction for prosthetic users using a visual analog scale from 0 to 100, where higher scores indicate more positive responses. Only certain subsets were used, including the ambulation subscale, satisfaction and safety questions, and utility questions. The hypothesis tested was that the new MPK has a 95% chance of not negatively affecting overall satisfaction. If scores in Visit 2 (with the investigational device) were higher than in Visit 1 (with the prescribed device), it would support the hypothesis. The confidence interval bars represented in graph were visually compared to the margin of non-inferiority. No further statistical analysis was done.
Time Frame: Baseline and After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
units on a scale
  Rheo Knee users: number analyzed (Participants) | 4
  Rheo Knee users | 2.6 [-6.2 to 11.5]
  Hydraulic users: number analyzed (Participants) | 6
  Hydraulic users | 7.4 [-9.1 to 23.8]
  All users | 5.5 [-3.4 to 14.3]

5. Primary Outcome: Change in Distance Walked During 2-Minute Walk Test (2MWT) From Baseline With Prescribed Device to After 4 Weeks of Investigational Device Use
Description: Average difference in distance walked in 2MWT with the new MPK compared to comparator (prescribed device) User walk for 2 minutes in their self selected walking speed on a 30 meter track.
  The hypothesis being tested is that the new MPK has a 95% probability of not negatively affecting the distance walked on 2MWT.
  For this hypothesis, if scores in visit 2 (subjects using the investigational device) were higher than in visit 1 (subjects using their prescribed device), the difference of Visit 2 - Visit 1 would be positive and would therefore support the corresponding hypothesis.
  The confidence interval bars represented in graph were visually compared to the margin of non-inferiority. No further statistical analysis was done.
Time Frame: Baseline and After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
meters
  Rheo Knee users: number analyzed (Participants) | 4
  Rheo Knee users | 2.43 [-6.1 to 11.0]
  Hydraulic users: number analyzed (Participants) | 6
  Hydraulic users | -1.8 [-6.1 to 2.4]
  All users | -0.1 [-3.6 to 3.3]

6. Primary Outcome: Change in Time for the Timed Up and Go Test (TUG) From Baseline With Prescribed Device to After 4 Weeks of Investigational Device Use
Description: The TUG test is a simple evaluative test used to measure functional mobility and assess fall risk. Reduction in time (measured in seconds) to complete indicates improvement in mobility. Average time needed to perform the TUG with the new MPK compared to comparator (prescribed device). The hypothesis being tested is that the new MPK has a 95% probability of not negatively affecting the time needed to complete the TUG. For this hypothesis, if the completion times of the TUG during the Visit 2 (subjects using the investigational device) were lower than the ones in Visit 1 (subjects using their prescribed device), the difference of Visit 2 - Visit 1 would be negative and would therefore support the corresponding hypothesis. The confidence interval bars represented in graph were visually compared to the margin of non-inferiority. No further statistical analysis was done.
Time Frame: Baseline and After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Mean (95% Confidence Interval); unit: time in seconds
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
time in seconds
  Rheo Knee users: number analyzed (Participants) | 4
  Rheo Knee users | -0.1 [-2.1 to 2.1]
  Hydraulic users: number analyzed (Participants) | 6
  Hydraulic users | -0.2 [-1.7 to 1.3]
  All users | -0.2 [-1.1 to 0.8]

7. Primary Outcome: Change in T-score for the Prosthetic Limb Users Survey of Mobility (PLUS-M) From Baseline With Prescribed Device to After 4 Weeks of Investigational Device Use
Description: Ability to ambulate over typical environmental obstacles is measured by the PLUS-M, using the T-score with the new MPK compared to the comparator (prescribed device). The PLUS-M is a self-report tool for assessing mobility in adults with lower limb amputation. The PLUS-M produces a T-score, which is standardized with a mean of 50 and a standard deviation of 10. Higher T-scores indicate greater mobility, with scores ranging from 17.5 to 76.6, based on responses to 44 questions. Only T-scores should be reported, as they are valid and comparable, unlike raw scores. The hypothesis being tested is that the new MPK has a 95% probability of not negatively affecting the PLUS-M score. If Visit 2 scores (using the investigational device) are higher than Visit 1 scores (using the prescribed device), the positive difference supports the hypothesis. The confidence interval bars represented in graph were visually compared to the margin of non-inferiority. No further statistical analysis was done.
Time Frame: Baseline and After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
T-score
  Rheo Knee users: number analyzed (Participants) | 4
  Rheo Knee users | 3.8 [-8.3 to 16.0]
  Hydraulic users: number analyzed (Participants) | 6
  Hydraulic users | 20.0 [-18.4 to 58.3]
  All users | 13.5 [-7.1 to 34.1]

8. Primary Outcome: Change in Activities-Specific Balance Confidence Score (ABC) From Baseline With Prescribed Device to After 4 Weeks of Investigational Device Use
Description: The ABC-scale is a 16-item questionnaire measuring confidence in performing ambulatory activities without falling, scored from 0 (no confidence) to 100 (full confidence). Cut-off scores define physical functioning: below 50% indicates low, 50-80% moderate, and above 80% high functioning. The hypothesis is that the new MPK has a 95% chance of not negatively impacting the ABC score. If Visit 2 scores (using the investigational device) exceed Visit 1 scores (using the prescribed device), it supports the hypothesis. Confidence interval bars in the graph were visually compared to the margin of non-inferiority, with no additional statistical analysis conducted.
Time Frame: Baseline and After 4 weeks of use
Population: 4 subjects had magnetorheological working MPK, 6 subjects had a hydraulic one.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Exploratory Testing of a New Prosthetic Knee
Number analyzed (Participants) | 10
score on a scale
  Rheo Knee users: number analyzed (Participants) | 4
  Rheo Knee users | 2.3 [-14.8 to 19.5]
  Hydraulic users: number analyzed (Participants) | 6
  Hydraulic users | 5.4 [-3.8 to 14.6]
  All users | 4.1 [-2.4 to 10.7]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Exploratory Testing of a New Prosthetic Knee
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exploratory Testing of a New Prosthetic Knee (N=11)
Unrelated issue on the residual limb (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT06748729/Prot_SAP_000.pdf